CLINICAL TRIAL: NCT02903849
Title: Using Self-Motivating Messages to Encourage People to Exercise More
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Hengchen Dai, Assistant Professor of Organizational Behavior, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016080382
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control (Experimental): On the 20th, 50th, and 90th day of the Challenge, Wellness Connection will email employees who participate in this survey. Employees will receive standard reminders generated by Wellness Connection.
  Interventions: Behavioral: Drafting Motivational Messages; Behavioral: Control Reminders
- Treatment (Experimental): On the 20th, 50th, and 90th day of the Challenge, Wellness Connection will email employees who participate in this survey. Employees will see the motivating messages they wrote at the beginning of the Challenge, in addition to Wellness Connection's standard reminders.
  Interventions: Behavioral: Drafting Motivational Messages; Behavioral: Treatment Reminders

INTERVENTIONS:
Behavioral: Drafting Motivational Messages — Write down three motivating messages
Behavioral: Control Reminders — Receive standard reminders at three points during the challenge
  Arms: Control
Behavioral: Treatment Reminders — Receive reminders containing the messages they leave themselves at three points during the challenge
  Arms: Treatment

SUMMARY:
The investigators are interested in using personalized, self-motivating messages to motivate people to exercise more.

DETAILED DESCRIPTION:
The investigators are interested in using personalized, self-motivating messages to motivate people to exercise more. Through a partnership with a university, the investigators are running a large-scale, randomized field controlled trial aimed at increasing exercise frequencies during a 100-day challenge. The primary purpose of this study is to test whether sending people motivating messages they wrote to themselves in the past can keep them engaged in the challenge and motivate them to exercise more frequently. One week into the challenge, employees who have signed up for the challenge will receive an email inviting them to participate in a short activity. Employees who click on the link will be directed to a survey. Once they finish reading the first introductory page and click "next", they will be randomly assigned to one of two groups. In the control group, employees will be encouraged to write down what they think will motivate them to walk more after 20, 50, and 90 days into the Challenge. These employees will receive standard reminders on the 20th, 50th, and 90th day of the challenge. In the treatment group, employees will be encouraged to write down motivating messages that they will receive on the 20th, 50th, and 90th day of the Challenge.

All employees who are exposed to either the control or the treatment condition will be included in the analysis.

The investigators plan to explore moderators based on (a) employees' demographics (age, gender, ethnicity, position), (b) employees' participation in previous challenges, and (c) employees' health condition and fitness level prior to the challenge (such as how actively they have been participating in other wellness activities, their health statistics).

ELIGIBILITY:
Inclusion Criteria:

* Employees who click on the link inviting them to participate in an activity and are assigned to either the treatment or control condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Activity Level | Through study completion, 100 days
  Number of steps taken each day, as recorded in participants' online portal.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | After the 100-day challenge ends
  Most recent BMI in pounds (weight) and inches (height) as entered by participant, an expected average of 2 months after study start. Obtaining the data is dependent on the ability to obtain the data from the online portal.
Cholesterol | After the 100-day challenge ends
  Most recent total, low, and high cholesterol levels in mg/dl as entered by participant, an expected average of 2 months after study start. Obtaining the data is dependent on the ability to obtain the data from the online portal.
Blood Pressure | After the 100-day challenge ends
  Most recent systolic and diastolic levels in mmHg as entered by participant, an expected average of 2 months after study start. Obtaining the data is dependent on the ability to obtain the data from the online portal.
Stress | After the 100-day challenge ends
  Most recent self-reported stress level on a 1-5 scale (with 1 indicating "Relaxed" and 5 indicating "Highly Stressed") as entered by participant, an expected average of 2 months after study start. Obtaining the data is dependent on the ability to obtain the data from the online portal.

CONTACTS AND LOCATIONS:
Overall Officials: Hengchen Dai, Ph.D, Principal Investigator — Washington University School of Medicine
Locations (1):
- Hengchen Dai, St Louis, Missouri, United States